CLINICAL TRIAL: NCT01608269
Title: Nucleoside Switch Pilot for Virologically Controlled HIV Subjects With Decreasing CD4 Cells Who Have Received TDF-based ARV Therapy
Acronym: EPZSwitch
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Therapeutic Concepts (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101-002
Record Dates: First submitted 2012-05-25; First posted 2012-05-31 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2012-05

CONDITIONS: HiV1- Positive
MeSH Terms: interventions — abacavir, lamivudine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ABC/3TC (Epzicom), NRTI (Other)
  Interventions: Drug: Abacavir/Lamivudine

INTERVENTIONS:
Drug: Abacavir/Lamivudine — one tablet once a day
  Other Names: ABC/3TC

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and antivira activity of Epzicom in virologically controlled HIV subjects.

DETAILED DESCRIPTION:
Utilizing the ABC/3TC FDC tablets as the NRTI backbone, this open label study will compare the safety and efficacy of ABC/3TC when used as replacement for subjects with suboptimal CD4- cells count who are receiving TDF/FTC. TYhis study will be conducted for 48 weeks in HIV infected, HLA*B5701 begative subjects who were initially suppressed on a HAART regiment that includes TDF/FTC QD.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 RNA ≤ 50 copies/mL by HIV-1 Ultrasensitive RNA, Quantitative.
* Treatment experienced subjects on virologically stable HAART regimen containing tenofovir-emtricitabine or tenofovir-lamivudine.
* Subject with CD4 cells that do not increase by 15% and/or that decrease by 15% over previous 12 months period.

  -≥ 18 years of age
* Cognitive ability to understand and provide written informed consent and willingness to participate in and comply with the study protocol
* Less than 7 days of prior ART with any licensed or investigational compound
* Patient does not currently have or has not been treated for an active opportunistic infection (OI) consistent with CDC definition (Appendix C) within 30 days of screening
* Vital signs, physical examination and laboratory results do not exhibit evidence of acute illness
* A female is eligible to enter and participate in this study if she is of:
* Non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal) or
* Child-bearing potential, has a negative serum pregnancy test at screen, and agrees to one of the following:
* Complete abstinence from intercourse from 2 weeks prior to administration of the study drug, throughout the study, and for at least 2 weeks after completion or premature discontinuation from the study to account for elimination of the investigational drug. Should a patient decide to become sexually active during the course of the study, she must be counseled and be willing to use one of the birth control methods listed below:
* Double barrier method (male condom/spermicide, male condom/diaphragm, diaphragm/spermicide)
* Any intrauterine device (IUD) with published data showing that the expected failure rate is <1% per year (not all IUDs meet this criterion)
* Sterilization (female patient or male partner of female patient)
* Any other methods with published data showing that the lowest expected failure rate for that method is <1% per year.

Exclusion Criteria:

* Patient with active AIDS-defining opportunistic infection or disease according to the 1993 CDC AIDS surveillance definition (Clinical Category C) in the 30 days prior to baseline and that, in the opinion of the investigator, would preclude the patient from participating in the study (See Appendix C).
* Patient who are HLA B5701 Positive
* Patient who are determined to have ≥2 thymidine analog mutations to RT
* History of active substance abuse, excluding cannabis, or psychiatric illness that, in the opinion of the investigator, would preclude compliance with protocol, dosing schedule and assessments.
* Patient is either pregnant at time of screening evaluation or breast-feeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-11; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Efficacy. | 1 years
  Proportion of patients with CD4 changes from baseline at week 24 and 48. Proportion of patients with plasma HIV-1 RNA <75 copies/mL at week 24 and 48

SECONDARY OUTCOMES:
Safety | 1 year
  Adverse events and treatment limiting toxicities at all time points.

CONTACTS AND LOCATIONS:
Locations (1):
- Therapeutic Concepts, PA, Houston, Texas, United States